CLINICAL TRIAL: NCT04962386
Title: Clinical Efficacy of Hormone Replacement Therapy in Treating Perimenopausal Women With Meibomian Gland Dysfunction
Brief Title: Clinical Efficacy of Hormone Replacement Therapy in Treating Perimenopausal Women With MGD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 研2019-363
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-06

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Hormone Replacement Therapy; Estradiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perimenopausal women who did not undergo HRT: Perimenopausal women who did not undergo HRT at baseline. And they did not receive any other drugs
  Interventions: Drug: Hormone replacement therapy
- Perimenopausal women who did undergo HRT: Perimenopausal women who did undergo HRT received estrogen-progesterone combination therapy packaged with estradiol tablets/estradiol and dynamic progesterone (Abbott Health Products BV. Weesp, The Netherlands).Take this medicine once a day. A course of treatment was defined as 28 days of continuous treatment.
  Interventions: Drug: Hormone replacement therapy

INTERVENTIONS:
Drug: Hormone replacement therapy — HRT women were treated with an estrogen-progesterone combination therapy packaged with estradiol tablets/estradiol and dynamic progesterone (Abbott Health Products BV, Weesp, the Netherlands).Take this medicine once a day.A course of treatment was defined as 28 days of continuous treatment.One white tablet containing 1mg of estradiol was taken daily for the first 14 days and one gray tablet containing 1mg of estradiol and 10 mg of dynamic progesterone was taken daily for the remaining 14 days.
  Other Names: Received estrogen-progesterone combination therapy packaged with estradiol tablets/estradiol and dynamic progesterone (Abbott Health Products BV, Weesp, The Netherlands)

SUMMARY:
This project aims to evaluate the possible relationship between MGD and HRT in perimenopausal women

DETAILED DESCRIPTION:
This project aims to: 1. Evaluate the possible relationship between MGD and HRT in perimenopausal women; 2. To explore the mechanism of HRT treatment on MGD through clinical trials;3. Optimize treatment methods by exploring the mechanism, and develop more personalized and systematic treatment plans for MDG patients in the perimenopausal period.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women who did not undergo HRT

Exclusion Criteria:

* (1) Patients who meet any of the following criteria will not be eligible for inclusion in the study: ① Unable or unwilling to sign a consent form, or unable to follow study procedures.

  (2) Have worn contact lenses in the past month, have had anterior segment surgery in the past 3 months, have a history of corneal refractive surgery, and have eye diseases other than dry eyes.Use of topical medicines other than eye lubricants in the past 3 months.Use of total body immunomodulators, tetracycline, or glucocorticoids in the past 3 months.Occlusion of lacrimal dots or eye trauma in the past 3 months.③ is pregnant, nursing or breastfeeding, or has received HRT treatment.

  ④ All patients with DE related diseases, such as diabetes mellitus, Sjogren syndrome, Stevens-Johnson syndrome.All participants were free of cancer, liver disease, kidney disease, stroke, transient cerebral ischemia, myocardial infarction, peptic ulcer, gout, or mental illness.Women who used anticoagulants, corticosteroids or vitamin A, vitamin E or beta-carotene were also excluded.

Ages: 25 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: MGD is a relatively new field of research in ophthalmology, so it has not been extensively studied up to now. However, MGD is believed to be a major cause of DE disease worldwide. It is estimated that MGD accounts for more than two-thirds of all DE cases. In one study, MGD accounted for 78 % of DE patients. The estimated incidence of MGD in Asian adults over 40 years of age ranges from 46.2% to 69.3%. Previous studies have shown that the production and stability of tears in postmenopausal women are reduced, and hormone replacement therapy can restore SLT values to the normal range. However, some studies have reported that women who receive HRT have a higher mortality rate than women who do not.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-03-06 (Estimated); Study Completion 2022-03-06 (Estimated)

PRIMARY OUTCOMES:
Tear secretion | 3 months
  After local anesthesia, a 35mm×5mm filter paper strip was placed longitudinally into the conjunctival sac of the lower eyelid. After 5 minutes, the length of the moist part was recorded. Less than 10mm was considered abnormal.

SECONDARY OUTCOMES:
Noninvasive tear break-up time test (NITBUT) | 3 months
  After fluorescein staining, patients were asked to close their eyes and measure the time until the first tear film break point appeared.The average of the three measurements was recorded and was considered abnormal for less than 10 seconds.
The scoring of corneal fluorescein staining | 3 months
  The cornea was divided into two groups on average. After staining, the upper, middle and lower corneal sites were recorded and the scores of each site were recorded.0= no punctate staining;1= less than half staining: 2= more than half staining;3= total staining;And the cumulative score (0-9 points) for each quadrant.CFS was assessed at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jin x ming, phd, Study Director — Second Affiliated Hospital of Zhejiang University Hospital
Locations (2):
- China (2):
  - Hangzhou Obstetrics and Gynecology Hospital, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Zhejiang University Hospital, Hangzhou

IPD SHARING:
Plan to Share IPD: No